CLINICAL TRIAL: NCT07398235
Title: A Qualitative Study to Explore the Barriers to Adoption of Clinical Decision Support Systems
Brief Title: A Qualitative Study Examining Clinical Decision Support System Adoption Among Hospital Clinicians
Acronym: CDSS-ADOPT
Status: Active, not recruiting | Type: Observational
Sponsor: Medway NHS Foundation Trust (Other)
Responsible Party: Principal Investigator, Saad Muhammad, Chief Investigator, Medway NHS Foundation Trust
Other Study IDs: 1366; IRAS ID: 365984 (Other: NHS Health Research Authority)
Record Dates: First submitted 2026-01-19; First posted 2026-02-09 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Clinical Decision Support System (CDSS)

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (7):
- FY1/2: Foundation Year 1 & 2 Doctors
  Interventions: Other: Semi-structured interview
- SHO: Senior House Officer level doctor above FY2 but below Registrar
  Interventions: Other: Semi-structured interview
- Registrar: Registrar level doctor
  Interventions: Other: Semi-structured interview
- Consultant: Consultant level doctor
  Interventions: Other: Semi-structured interview
- Physician Assistant: Physician Assistant clinician
  Interventions: Other: Semi-structured interview
- ANP: Advanced Nurse Practitioner
  Interventions: Other: Semi-structured interview
- CSW: Clinical Support Worker
  Interventions: Other: Semi-structured interview

INTERVENTIONS:
Other: Semi-structured interview — A 20-30 minute semi-structured interview using the pre-defined topic sheet

SUMMARY:
A Qualitative Study to Explore the Barriers to Adoption of Clinical Decision Support Systems

DETAILED DESCRIPTION:
Qualitative study looking at clinical decision support system adoption among clinicians in a district general hospital. This will involve semi-structured interviews of various clinical staff in the emergency department, looking at work-habits regarding clinical decision support tool use.

ELIGIBILITY:
Inclusion Criteria:

* Employed by Medway NHS Foundation Trust at the time of recruitment
* Working clinically within the Emergency Department
* Clinical grade of FY1, FY2, SHO/CTF, SAS/Registrar, Consultant, Nurse, Advanced Clinical practitioner, Physician Assistant, or Clinical Support Worker
* Involved in the assessment and management of adult emergency department patients
* Have routine access to the Trust electronic patient record system (Sunrise EPR) during clinical duties
* Able to provide informed consent to participate
* Aged 18 years or older

Exclusion Criteria:

* Bank, agency, or locum staff who are not permanently or regularly employed by the department.
* Staff currently on leave, secondment, or not actively practising in the ED during the data collection period.
* Clinicians currently involved in the design, management, or evaluation of the CDSS system under study.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Hospital clinicians employed by Medway NHS Foundation Trust
Sampling Method: Non-Probability Sample
Enrollment: 12 (Estimated)
Dates: Start 2026-01-10 (Actual); Primary Completion 2026-01-31 (Actual); Study Completion 2026-02-21 (Estimated)

PRIMARY OUTCOMES:
Saturation of Themes Related to Barriers to CDSS Adoption | The study ran between 10th January 2026 until 31 January 2026. The study was considered complete once all planned participant interviews have been conducted or recruitment has formally ceased following achievement of data saturation.
  The primary outcome examines the barriers to clinical decision support system adoption, such as hardware issues, governance concerns, user-interface problems, and trusted information. These themes will be examined during interviews with open-ended questions to allow user experiences to be recorded.
  This study will use purposive sampling with maximum variation to ensure representation across key categories of Emergency Department clinicians who use clinical decision support systems (CDSS). Participants will be selected to capture a range of roles and experiences, including Advanced Clinical Practitioners (ACPs), Physician Associates (PAs), Clinical Support Workers (CSWs), nurses, and doctors at different levels (Foundation Year 1-2, Senior House Officers, Registrars, and Consultants). Recruitment will continue until data saturation of themes related to CDSS adoption is achieved within and across these categories, anticipated at approximately one to two participants per role group.

CONTACTS AND LOCATIONS:
Locations (1):
- Medway NHS Foundation Trust, Gillingham, Kent, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mebrahtu TF, Skyrme S, Randell R, Keenan AM, Bloor K, Yang H, Andre D, Ledward A, King H, Thompson C. Effects of computerised clinical decision support systems (CDSS) on nursing and allied health professional performance and patient outcomes: a systematic review of experimental and observational studies. BMJ Open. 2021 Dec 15;11(12):e053886. doi: 10.1136/bmjopen-2021-053886. PMID 34911719
- [Background] Meunier PY, Raynaud C, Guimaraes E, Gueyffier F, Letrilliart L. Barriers and Facilitators to the Use of Clinical Decision Support Systems in Primary Care: A Mixed-Methods Systematic Review. Ann Fam Med. 2023 Jan-Feb;21(1):57-69. doi: 10.1370/afm.2908. PMID 36690490
- [Background] Chen W, O'Bryan CM, Gorham G, Howard K, Balasubramanya B, Coffey P, Abeyaratne A, Cass A. Barriers and enablers to implementing and using clinical decision support systems for chronic diseases: a qualitative systematic review and meta-aggregation. Implement Sci Commun. 2022 Jul 28;3(1):81. doi: 10.1186/s43058-022-00326-x. PMID 35902894
- [Background] Liberati EG, Ruggiero F, Galuppo L, Gorli M, Gonzalez-Lorenzo M, Maraldi M, Ruggieri P, Polo Friz H, Scaratti G, Kwag KH, Vespignani R, Moja L. What hinders the uptake of computerized decision support systems in hospitals? A qualitative study and framework for implementation. Implement Sci. 2017 Sep 15;12(1):113. doi: 10.1186/s13012-017-0644-2. PMID 28915822
- [Background] Pardo GI, Renner RP. The telescoped overdenture: advantages and limitations. J Am Dent Assoc. 1980 Dec;101(6):932-4. doi: 10.14219/jada.archive.1980.0457. PMID 7005290
- See also: 10 Year Health Plan for England (Department of Health and Social Care) — https://www.gov.uk/government/publications/10-year-health-plan-for-england-fit-for-the-future
- See also: Independent Investigation of the NHS in England (Department of Health and Social Care) — https://www.gov.uk/government/publications/independent-investigation-of-the-nhs-in-england
- See also: Supporting clinical decisions with health information technology: An implementation guide for clinical decision support systems (NHS England) — https://www.england.nhs.uk/long-read/supporting-clinical-decisions-with-health-information-technology
- See also: NASSS-CAT Toolkit (Thrive by Design) — https://www.thrivebydesign.org.uk/our-learning/nasss-cat-toolkit

DOCUMENTS (2):
  • Study Protocol (2026-01-06): https://cdn.clinicaltrials.gov/large-docs/35/NCT07398235/Prot_000.pdf
  • Informed Consent Form (2026-01-06): https://cdn.clinicaltrials.gov/large-docs/35/NCT07398235/ICF_001.pdf